CLINICAL TRIAL: NCT01533948
Title: Predictive Markers of Response in a Phase II Trial of Axitinib in Advanced Melanoma
Brief Title: Axitinib in Treating Patients With Melanoma That is Metastatic or Cannot Be Removed by Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 197811; NCI-2011-03037 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 197811 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2012-01-18; First posted 2012-02-16 (Estimated); Results first posted 2018-05-09 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Extraocular Extension Melanoma; Metastatic Intraocular Melanoma; Recurrent Intraocular Melanoma; Recurrent Melanoma; Stage IIIA Intraocular Melanoma; Stage IIIA Melanoma; Stage IIIB Intraocular Melanoma; Stage IIIB Melanoma; Stage IIIC Intraocular Melanoma; Stage IIIC Melanoma; Stage IV Intraocular Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (axitinib) (Experimental): Patients receive axitinib PO BID. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: axitinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: axitinib — Given PO
  Other Names: AG-013736; Inlyta
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well axitinib works in treating patients with melanoma that has spread to other places in the body or cannot be removed by surgery. Axitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall response rate (ORR) to axitinib in advanced melanoma. This will be assessed using the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1.

SECONDARY OBJECTIVES:

I. Evaluate toxicity of axitinib as a single agent. II. Determine progression-free survival and overall survival. III. Explore the utility of 3'-deoxy-3'-[18F] fluorothymidine-labeled positron emission tomography (FLT-PET) as a predictive marker for response and compare to standard radiographic imaging.

TERTIARY OBJECTIVES:

I. Examine the prognostic and predictive significance of circulating melanoma tumor cells.

II. To examine whether functionally relevant polymorphisms in axitinib-related genes (vascular endothelial growth factor receptor [VEGFR] 1, VEGFR2 and VEGFR3) correlate with efficacy and toxicity of axitinib in advanced melanoma.

OUTLINE:

Patients receive axitinib orally (PO) twice daily (BID). Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven melanoma (including uveal) that is advanced (metastatic) or unresectable
* Measurable disease
* No more than two prior regimens (0-2) of systemic therapy for metastatic or recurrent disease; therapy (systemic or radiotherapy) administered in the neo-adjuvant or adjuvant setting for previously localized disease is permitted, provided it was completed more than 3 months prior to enrollment; palliative radiotherapy is permitted provided it is completed >= 2 weeks prior to study therapy initiation and there is at least one measurable lesion outside the radiation field; at least 2 weeks since the end of prior systemic treatment, radiotherapy, or surgical procedure with resolution of all treatment-related toxicity to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 grade =< 1 or back to baseline except for alopecia or hypothyroidism
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Life expectancy >= 12 weeks
* Absolute neutrophil count (ANC) >= 1500 cells/mm^3
* Platelets >= 75,000 cells/mm^3
* Hemoglobin >= 9.0 g/dL
* Creatinine =< 1.5 X upper limit normal (ULN) or calculated creatinine clearance >= 60 mL/min
* Bilirubin =< 1.5 X ULN
* Transaminase =< 2.5 X ULN (for documented liver metastases, transaminase up to 5 X ULN is permitted)
* Random urinary protein/creatinine ratio < 2
* Have the ability to swallow and retain oral medication
* No evidence of preexisting uncontrolled hypertension as documented by 2 baseline blood pressure readings taken at least 1 hour apart; the baseline systolic blood pressure readings must be =< 140 mm Hg, and the baseline diastolic blood pressure readings must be =< 90 mm Hg; patients whose hypertension is controlled by antihypertensive therapies are eligible
* Women of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to treatment
* Patients of child-bearing potential must agree to use acceptable contraceptive methods (e.g., double barrier) during treatment and for 6 months following completion of study treatment
* Patient or legal representative must understand the investigational nature of this study and sign an Institutional Review Board (IRB) approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Prior anti-angiogenic therapy
* Major surgery < 4 weeks or radiation therapy < 2 weeks of starting the study treatment; prior palliative radiotherapy to metastatic lesion(s) is permitted, provided there is at least 1 measurable lesion that has not been irradiated
* Significant history of bleeding events (e.g., hemoptysis, grade 3 or grade 4 gross hematuria) within 6 months prior to registration
* Presence of serious non-healing wounds, ulcers (including gastro-intestinal) and bone fractures
* Gastrointestinal abnormalities including:

  * Inability to take oral medication
  * Requirement for intravenous alimentation
  * Prior surgical procedures affecting absorption including total gastric resection; segmental small bowel or colon resection is permitted
  * Treatment for active peptic ulcer disease in the past 6 months
  * Active gastrointestinal bleeding, unrelated to cancer, as evidenced by hematemesis, hematochezia or melena in the past 6 months without evidence of resolution documented by endoscopy or colonoscopy
  * Malabsorption syndromes
  * History of gastrointestinal (GI) perforation within prior 12 months
* Current use or anticipated need for treatment with drugs that are known potent cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors (i.e., grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, erythromycin, telithromycin, clarithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir and delavirdine)
* Current use or anticipated need for treatment with drugs that are known CYP3A4 or cytochrome P450, family 1, subfamily A, polypeptide 2 (CYP1A2) inducers (i.e., carbamazepine, dexamethasone, felbamate, omeprazole, phenobarbital, phenytoin, amobarbital, nevirapine, primidone, rifabutin, rifampin, and St. John's wort)
* Requirement of therapeutic anticoagulant therapy with oral vitamin K antagonists; low-dose anticoagulants for maintenance of patency of central venous access devise or prevention of deep venous thrombosis is allowed; therapeutic use of low molecular weight heparin (or similar parenteral drug) for venous-thromboembolic disease is allowed
* Active seizure disorder or evidence of untreated brain metastases, spinal cord compression, or carcinomatous meningitis; patients with brain metastases that have been stable for >= 4 weeks by radiographic documentation following definitive therapy will be permitted provided this is not the only site of metastatic disease
* Arterial thrombotic events within 6 months of registration, including myocardial infarction, unstable angina or angina requiring medical or surgical intervention in the past 6 months, coronary/peripheral artery bypass graft, cerebrovascular accident, transient ischemic attack and clinically significant peripheral vascular disease (i.e., claudication on less than 1 block)
* Current congestive heart failure (New York Heart Association [NYHA] class II, III or IV)
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness
* History of a malignancy except those treated with curative intent for skin cancer (other than melanoma), in-situ breast or in-situ cervical cancer, or those treated with curative intent for any other cancer with no evidence of disease for 3 years
* Female patients who are pregnant or lactating
* Received an investigational agent within 30 days prior to enrollment
* A serious uncontrolled medical disorder or active infection that would impair their ability to receive study treatment
* Any condition which in the investigator's opinion would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matuesz Opyrchal, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Axitinib): Patients receive axitinib PO BID. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  axitinib: Given PO
  The starting dose for axitinib is 5 mg taken orally twice daily with food. Axitinib will be taken beginning on Day 1 of the study and taken approximately 12 hours apart continuous dosing.
  Dose Level Dose Dispensed As
  * 2: 10 mg PO BID 2 X 5 mg tablets BID
  * 1: 7 mg PO BID 1 X 5 mg tablet BID + 2 X 1 mg tablets BID 0: (Starting Dose) 5 mg PO BID 1 X 5 mg tablet BID
    * 1: 3 mg PO BID 3 X 1 mg tablets BID
    * 2: 2 mg PO BID 2 X 1 mg tablets BID
Period: Overall Study
Arm/Group | Treatment (Axitinib)
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Treatment (Axitinib)
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Complete Response + Partial Response) to Axitinib as Assessed Using RECIST Version 1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 30 days
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Axitinib)
Number analyzed (Participants) | 25
percentage of participants | 12 [3 to 31]

2. Secondary Outcome: Number of Patients That Experienced at Least One Grade 3 Adverse Event
Description: Number of patients that experienced at least one grade 3 toxicity regardless of attribution. Incidence of toxicity of axitinib as a single agent as assessed by the severity of adverse effects by NCI CTCAE version 4. Please refer to the adverse event reporting for more detail.
Time Frame: Up to 30 days
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Axitinib)
Number analyzed (Participants) | 25
Participants | 12

3. Secondary Outcome: Median Progression-free Survival (PFS)
Description: The distribution will be described using Kaplan-Meier and proportional hazards methods. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From the date of study enrollment to the first observation of progressive disease or death within 30 days after last dose of study drug
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Axitinib)
Number analyzed (Participants) | 25
months | 2.1 [1.8 to 4.5]

4. Secondary Outcome: Median Overall Survival (OS)
Description: The distribution will be described using Kaplan-Meier and proportional hazards methods.
Time Frame: From the date of study enrollment to the time of death within 30 days after last dose of study drug
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Axitinib)
Number analyzed (Participants) | 25
months | 7.4 [5.5 to 18.3]

5. Secondary Outcome: The Baseline Circulative Tumor Cells Value of Responders
Description: The baseline Circulative tumor Cells values of patients with response to treatment per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. CTC were evaluated at baseline, response was assessed up to 30 days.
Time Frame: Baseline
Population: All treated and eligible patients that responded
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Treatment (Axitinib)
Number analyzed (Participants) | 3
cells/mm^3 | 0 (0)

ADVERSE EVENTS:
Arm/Group | Treatment (Axitinib)
Serious Adverse Events (participants affected / at risk) | 8/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Axitinib) (N=25)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (19)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Ascites (Gastrointestinal disorders) | 1 (6)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (8)
Small intestinal perforation (Gastrointestinal disorders) | 1 (6)
Death (General disorders) | 1 (13)
Sepsis (Infections and infestations) | 1 (17)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (28)
Haemorrhage intracranial (Nervous system disorders) | 1 (37)
Confusional state (Psychiatric disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Axitinib) (N=25)
Anaemia (Blood and lymphatic system disorders) | 1 (22)
Lymph node pain (Blood and lymphatic system disorders) | 1 (2)
Hyperthyroidism (Endocrine disorders) | 1 (17)
Hypothyroidism (Endocrine disorders) | 9 (13)
Abdominal distension (Gastrointestinal disorders) | 1 (24)
Abdominal pain (Gastrointestinal disorders) | 5 (29)
Abdominal pain lower (Gastrointestinal disorders) | 1 (7)
Abdominal pain upper (Gastrointestinal disorders) | 1 (35)
Constipation (Gastrointestinal disorders) | 4 (9)
Dental caries (Gastrointestinal disorders) | 1 (14)
Diarrhoea (Gastrointestinal disorders) | 10 (54)
Dry mouth (Gastrointestinal disorders) | 2 (13)
Dyspepsia (Gastrointestinal disorders) | 2 (31)
Flatulence (Gastrointestinal disorders) | 1 (18)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (16)
Nausea (Gastrointestinal disorders) | 5 (11)
Oesophageal pain (Gastrointestinal disorders) | 1 (7)
Paraesthesia oral (Gastrointestinal disorders) | 3 (27)
Stomatitis (Gastrointestinal disorders) | 8 (19)
Vomiting (Gastrointestinal disorders) | 2 (20)
Asthenia (General disorders) | 1 (22)
Fatigue (General disorders) | 15 (26)
Mucosal inflammation (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 1 (78)
Bacteraemia (Infections and infestations) | 1 (10)
Gastrointestinal infection (Infections and infestations) | 1 (5)
Infusion site infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (15)
Sinusitis (Infections and infestations) | 1 (8)
Tooth infection (Infections and infestations) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (4)
Limb injury (Injury, poisoning and procedural complications) | 1 (14)
Alanine aminotransferase increased (Investigations) | 3 (15)
Aspartate aminotransferase increased (Investigations) | 9 (14)
Blood alkaline phosphatase increased (Investigations) | 2 (19)
Blood thyroid stimulating hormone increased (Investigations) | 1 (12)
Haemoglobin decreased (Investigations) | 1 (10)
Lymphocyte count decreased (Investigations) | 6 (16)
Platelet count decreased (Investigations) | 1 (6)
Weight decreased (Investigations) | 6 (13)
Cachexia (Metabolism and nutrition disorders) | 1 (6)
Decreased appetite (Metabolism and nutrition disorders) | 7 (13)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (4)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (10)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (57)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (32)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (22)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (8)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (18)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (18)
Dizziness (Nervous system disorders) | 1 (17)
Dysgeusia (Nervous system disorders) | 5 (21)
Headache (Nervous system disorders) | 5 (37)
Neuralgia (Nervous system disorders) | 1 (8)
Sinus headache (Nervous system disorders) | 1 (4)
Anxiety (Psychiatric disorders) | 4 (30)
Confusional state (Psychiatric disorders) | 1 (15)
Depression (Psychiatric disorders) | 2 (31)
Insomnia (Psychiatric disorders) | 2 (17)
Haematuria (Renal and urinary disorders) | 1 (16)
Nocturia (Renal and urinary disorders) | 1 (5)
Proteinuria (Renal and urinary disorders) | 2 (4)
Renal failure acute (Renal and urinary disorders) | 1 (28)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (20)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 14 (18)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (31)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (9)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (14)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (13)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (11)
Erythema (Skin and subcutaneous tissue disorders) | 1 (32)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (11)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 10 (18)
Rash (Skin and subcutaneous tissue disorders) | 2 (36)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (9)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (38)
Hypertension (Vascular disorders) | 10 (35)
Hypotension (Vascular disorders) | 3 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes